CLINICAL TRIAL: NCT06048653
Title: Effect of Non-invasive Vagus Nerve Stimulation on Cognitive Functions in Diabetic Polyneuropathy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: heba ahmed khalifa (Other)
Responsible Party: Sponsor-Investigator, heba ahmed khalifa, Ass. Prof. Dr of Physical therapy for Neurology, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003942
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: vagus nerve stimulation; cognitive functions
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The control group (GI) will receive a computer based cognitive rehabilitation program (Rehacom system); and the study group (GII) will receive the same program as (GI) in addition to Vagus nerve stimulation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): The control group (GI) will receive a computer based cognitive rehabilitation program (Rehacom system)
  Interventions: Other: A computer based cognitive rehabilitation program (Rehacom system)
- study group (Experimental): The study group (GII) will receive a computer based cognitive rehabilitation program (Rehacom system) in addition to Vagus nerve stimulation.
  Interventions: Other: A computer based cognitive rehabilitation program (Rehacom system); Device: Vagus nerve stimulation

INTERVENTIONS:
Other: A computer based cognitive rehabilitation program (Rehacom system) — Rehacom cognitive rehabilitation software will be used to treat the cognitive dysfunction
  * Patients will receive training for four weeks, two sessions per week.
  * Each patient will assume a comfortable sitting position on a chair in front of the screen.
  * A report will be generated at the end of the session. It will be used for follow up.
  * Session duration will range from 45 to 60 min. including rest period.
Device: Vagus nerve stimulation — stimulation will be applied on cymba conchae of left external ear. A stimulation of frequency of 20 Hz, pulse width of 200 - 300 Ms and intensity of 0.5 mA. The stimulation will be on for 30 s and off for 48 s.The stimulus duration will range from 20 to 40 min.
  Arms: study group

SUMMARY:
Diabetic peripheral neuropathy (DPN) occurs due to long standing hyperglycemia and associated metabolic derangements. Cognitive impairment is a common complication in diabetes mellitus. It is associated with a faster rate of cognitive decline.

DETAILED DESCRIPTION:
This research aims to

* determine the effect of non-invasive Vagus nerve stimulation on cognitive functions in diabetic peripheral neuropathy.
* investigate the correlation between cognitive function and severity of diabetic neuropathy.
* investigate the correlation between cognitive function and quality of life in diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetic polyneuropathy
* Female patients.
* age ranges from 40 to 55 years old.
* Duration of diabetic illness started since at least three years.
* Patients with mild to moderate neuropathy according to Toronto clinical neuropathy score
* Patients with cognitive function ranges from 24 - 15 score according to Mini mental state examination
* Patients with HbA1c ranges from seven to nine score.
* Ambulant patients with or without walking aids.
* Medically and psychologically stable patients without cardiac problems, confirmed by Electro Cardiogram (ECG).
* able to understand instructions.

Exclusion Criteria:

* Type I diabetes mellitus.
* Severe visual, verbal or acoustic impairments.
* Sever cognitive dysfunctions or that caused by other cause rather than diabetes mellitus.
* Polyneuropathy caused by other cause rather than diabetes mellitus.
* Other neurological problem as stroke.
* Cardiovascular problems.
* Metallic implants
* Illiterate patients.
* Uncooperative patients.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Diabetic polyneuropathy female patients
Enrollment: 40 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Attention/ concentration score | at baseline
  Rehacom will be used to assess score of attention/ concentration domain of cognitive function
Attention/ concentration score | post intervention (after one month)
  Rehacom will be used to assess score of attention/ concentration domain of cognitive function
working memory score | at baseline
  Rehacom will be used to assess score of working memory domain of cognitive function
working memory score | post intervention (after one month)
  Rehacom will be used to assess score of working memory domain of cognitive function
Executive function score | at baseline
  Rehacom will be used to assess score of executive function domain of cognitive function
Executive function | post intervention (after one month)
  Rehacom will be used to assess score of executive function domain of cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Moshera Darwish, Prof. Dr, Principal Investigator — Professor of Physical therapy for Neurology
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awad N, Gagnon M, Messier C. The relationship between impaired glucose tolerance, type 2 diabetes, and cognitive function. J Clin Exp Neuropsychol. 2004 Nov;26(8):1044-80. doi: 10.1080/13803390490514875. PMID 15590460
- [Background] Broncel A, Bocian R, Klos-Wojtczak P, Kulbat-Warycha K, Konopacki J. Vagal nerve stimulation as a promising tool in the improvement of cognitive disorders. Brain Res Bull. 2020 Feb;155:37-47. doi: 10.1016/j.brainresbull.2019.11.011. Epub 2019 Nov 29. PMID 31790720
- [Derived] Darwish MH, El-Tamawy MS, Alhirsan SM, El-Anany M, Khalifa HA. Effect of Trans-Auricular Vagal Nerve Stimulation on Cognitive Functions in Diabetic Polyneuropathy Patients. Physiother Res Int. 2025 Apr;30(2):e70063. doi: 10.1002/pri.70063. PMID 40285458